CLINICAL TRIAL: NCT07020325
Title: Comparative Analysis of Bipolar Enucleation of the Prostate Using Different Commercial Types of Electrodes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Mohamed Kamal Omar, Clinical Professor of Urology in Menoufia University, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2/2025 Urol
Record Dates: First submitted 2025-03-25; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Bipolar Enucleation of the Prostate

STUDY DESIGN:
Intervention Model Description: This study follows a parallel design, where participants are randomly assigned to one of four intervention groups. Each group receives treatment with a specific type of commercial bipolar electrode. The study aims to assess differences in efficacy, safety, learning curve, and cost-effectiveness across the four electrode types. The surgical technique is standardized across all centers to minimize variability, and data collection is blinded to ensure objective analysis.
Who Masked: Outcomes Assessor
Masking Description: Data collection and analysis will be conducted by blinded investigators to minimize bias. While surgeons performing the procedures will be aware of the electrode type used, the outcomes assessors evaluating postoperative results will remain blinded to ensure objective assessment of efficacy, safety, complications, and cost-effectiveness.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Bipolar Enucleation Using Electrode A (Company X) (Experimental): Participants will undergo prostate enucleation using Electrode A for BPH treatment.
  Interventions: Procedure: Bipolar Enucleation of the Prostate; Device: Bipolar electrode From Wolf company
- Bipolar Enucleation Using Electrode B (Company Y) (Experimental): Participants will undergo prostate enucleation using Electrode B for BPH treatment.
  Interventions: Procedure: Bipolar Enucleation of the Prostate; Device: Bipolar electrode From Storz company
- Bipolar Enucleation Using Electrode C (Company W) (Experimental): Bipolar Enucleation Using Electrode C (Company W)
  Interventions: Procedure: Bipolar Enucleation of the Prostate; Device: Bipolar electrode From Olympus company
- Bipolar Enucleation Using Electrode D (Company Z) (Experimental): Bipolar Enucleation Using Electrode D (Company Z)
  Interventions: Procedure: Bipolar Enucleation of the Prostate; Device: Bipolar electrode From Lamidey company

INTERVENTIONS:
Procedure: Bipolar Enucleation of the Prostate — Bipolar enucleation of the prostate involves the removal of prostate tissue using a bipolar electrode. This procedure is performed for patients with benign prostatic hyperplasia (BPH), with different electrode types used for comparison in this study
Device: Bipolar electrode From Wolf company — This study involves bipolar transurethral resection of the prostate (TURP) using four different bipolar electrosurgical systems, each provided by a distinct manufacturer. The aim is to evaluate and compare the efficacy, safety, and clinical outcomes associated with each system.
  Arms: Bipolar Enucleation Using Electrode A (Company X)
Device: Bipolar electrode From Storz company — This study involves bipolar transurethral resection of the prostate (TURP) using four different bipolar electrosurgical systems, each provided by a distinct manufacturer. The aim is to evaluate and compare the efficacy, safety, and clinical outcomes associated with each system.
  Arms: Bipolar Enucleation Using Electrode B (Company Y)
Device: Bipolar electrode From Olympus company — This study involves bipolar transurethral resection of the prostate (TURP) using four different bipolar electrosurgical systems, each provided by a distinct manufacturer. The aim is to evaluate and compare the efficacy, safety, and clinical outcomes associated with each system.
  Arms: Bipolar Enucleation Using Electrode C (Company W)
Device: Bipolar electrode From Lamidey company — This study involves bipolar transurethral resection of the prostate (TURP) using four different bipolar electrosurgical systems, each provided by a distinct manufacturer. The aim is to evaluate and compare the efficacy, safety, and clinical outcomes associated with each system.
  Arms: Bipolar Enucleation Using Electrode D (Company Z)

SUMMARY:
The goal of this randomized, prospective, multicenter clinical trial is to compare the enucleation efficacy of prostate enucleation using different commercial bipolar electrodes in male patients aged ≥50 years diagnosed with benign prostatic hyperplasia (BPH). The main questions it aims to answer are:

Which bipolar electrode provides the most effective enucleation?

What are the safety and postoperative outcomes of different bipolar electrodes?

What are the intraoperative and postoperative complication rates for each electrode type?

How does the learning curve differ among different electrode types?

What is the cost-effectiveness of each electrode?

Researchers will compare four groups, each assigned a different commercial bipolar electrode (Electrode A, B, C, or D), to determine differences in efficacy, safety, and cost-effectiveness.

Participants will:

Undergo bipolar enucleation of the prostate performed by experienced surgeons.

Be randomized into one of four groups based on the electrode used.

Follow a standardized surgical technique across all centres.

Be monitored for intraoperative and postoperative outcomes over a 6-month follow-up period.

Data collection and analysis will be conducted by blinded investigators to ensure unbiased results.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥50 years
* Diagnosed with moderate to severe LUTS due to BPH.
* Prostate size ≥40 g based on transrectal ultrasound (TRUS) or MRI.
* Ability to provide informed consent.

Exclusion Criteria:

* Prostate cancer.
* Urethral stricture disease.
* Patients with severe cardiac comorbidities or bleeding disorders.
* Patients on anticoagulation therapy.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-02-10 (Estimated); Study Completion 2026-03-10 (Estimated)

PRIMARY OUTCOMES:
Enucleation Efficiency (g/min) of Different Bipolar Electrodes | Time Frame: Intraoperative
  Enucleation efficiency will be calculated by dividing the enucleated tissue weight (grams) by the total enucleation time (minutes), providing a g/min value. This metric reflects the technical efficacy of the bipolar enucleation electrode in prostate tissue removal. Data will be compared across the four bipolar systems used in the study.

SECONDARY OUTCOMES:
Perioperative Safety: Incidence of Adverse Events (Clavien-Dindo Classification) | Time Frame: Intraoperative and up to 30 days postoperative
  Complications will be recorded and graded according to the Clavien-Dindo classification system. Events include, but are not limited to, bleeding requiring transfusion, urinary retention, infection, bladder injury, and incontinence. The frequency and severity of complications will be analyzed and compared between devices.
  Unit of Measure: Number of adverse events per Clavien-Dindo grade.
Change in International Prostate Symptom Score (IPSS) | Time Frame: Preoperative baseline, and at 6 weeks, 3 months, and 6 months postoperative
  Description: Change from baseline in patient-reported urinary symptoms as measured by the International Prostate Symptom Score (IPSS) to evaluate symptom improvement after bipolar enucleation.
  Unit of Measure: IPSS score (0-35)
Change in Maximum Flow Rate (Qmax) | Time Frame: Preoperative baseline, 6 weeks, 3 months, and 6 months postoperative
  Description: Change from baseline in maximum urinary flow rate to assess improvement in urinary flow after bipolar enucleation.
  Unit of Measure: mL/second
Change in Post-Void Residual Volume (PVR) | Time Frame: Preoperative baseline, 6 weeks, 3 months, and 6 months postoperative
  Description: Change from baseline in post-void residual urine volume to evaluate bladder emptying efficiency after bipolar enucleation.
  Unit of Measure: milliliters (mL)
Learning Curve Assessment Based on Enucleation Time Over Consecutive Cases | During 12-month recruitment/study period
  Surgeon learning curve will be assessed by measuring enucleation time (in minutes) across consecutive cases for each bipolar system. The trend in time reduction will be analyzed to evaluate the learning trajectory.
  Unit of Measure: Enucleation time in minutes per case
Cost-Effectiveness: Total Procedure and Postoperative Cost per Patient | Time Frame: From procedure day to end of 6-month follow-up
  Total cost per patient will be calculated by summing surgical device costs, operating room time, length of hospital stay, and postoperative care costs (including catheter duration, readmissions, and complication-related expenses).
  Unit of Measure: Cost in local currency (e.g., Euros or USD)